CLINICAL TRIAL: NCT07395102
Title: Effectiveness of Thread-Embedding Acupuncture at EX-B2 on the Oswestry Disability Index and Finger-to-Floor Distance in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Desi Recsanti, Principal Investigator, Faculty of Medicine, Universitas Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-12-1949
Record Dates: First submitted 2026-01-25; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups:
  Thread Embedding Acupuncture (TEA) group
  Sham Thread Embedding Acupuncture (Control) group
  Both groups will receive procedures with identical appearance and schedule. The intervention group will receive implantation of absorbable polydioxanone (PDO) threads at EX-B2 acupuncture points, while the control group will receive a sham procedure without thread implantation. Participants will be followed for 8 weeks after the intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to group allocation. The sham procedure will be designed to be visually and procedurally similar to the active thread embedding acupuncture intervention. Outcome assessors will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Thread Embedding Acupuncture (TEA) (Experimental): Participants in this group will receive thread embedding acupuncture using absorbable polydioxanone (PDO) threads implanted bilaterally at EX-B2 acupuncture points corresponding to the lumbar vertebral segments. The procedure will be performed only once weekly at week 0. This intervention is intended to provide continuous stimulation of acupuncture points to reduce disability and improve lumbar flexibility in patients with chronic low back pain.
  Interventions: Device: Thread Embedding Acupuncture
- Control Group - Sham Thread Embedding Acupuncture (Sham Comparator): Participants in the control group will receive a sham thread embedding acupuncture procedure that mimics the intervention in terms of patient positioning, skin preparation, and needle insertion technique, but without implantation of polydioxanone (PDO) threads. No absorbable thread will be left in the tissue. The procedure will be performed only once weekly at week 0. This group serves as a placebo control to evaluate the specific effects of thread embedding acupuncture beyond nonspecific procedural effects.
  Interventions: Device: Sham Thread Embedding Acupuncture

INTERVENTIONS:
Device: Thread Embedding Acupuncture — Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups. The assigned procedures will be administered once, and outcomes will be evaluated over an 8-week follow-up period.
  Arms: Intervention Group - Thread Embedding Acupuncture (TEA)
Device: Sham Thread Embedding Acupuncture — Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups. The assigned procedures will be administered once, and outcomes will be evaluated over an 8-week follow-up period.
  Arms: Control Group - Sham Thread Embedding Acupuncture

SUMMARY:
Chronic low back pain (CLBP) is a leading cause of disability worldwide and significantly impairs functional capacity and quality of life. Non-pharmacological therapies are recommended as first-line management, and acupuncture has demonstrated potential benefits in reducing pain and disability. Thread embedding acupuncture (TEA) is a modified acupuncture technique that provides prolonged stimulation through the implantation of absorbable polydioxanone (PDO) threads at acupuncture points.

This randomized controlled trial aims to evaluate the effectiveness of TEA at the EX-B2 points compared with sham TEA in improving disability and lumbar flexibility in patients with chronic non-specific low back pain. Disability will be assessed using the Oswestry Disability Index (ODI), and lumbar flexibility will be measured using the Finger-to-Floor Distance (FFD) test over an 8-week follow-up period.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a major contributor to global disability and reduced functional performance. Conventional management such as analgesics and physiotherapy often provides limited long-term functional improvement. Acupuncture has been recommended as a non-pharmacological treatment option for CLBP, and evidence suggests it can reduce pain and disability.

Thread embedding acupuncture (TEA) is a modified acupuncture technique in which absorbable medical threads are implanted into specific acupuncture points, providing continuous stimulation over several weeks. This prolonged stimulation is believed to enhance neuromodulation, improve local microcirculation, and promote tissue repair, potentially leading to sustained clinical benefits.

The EX-B2 points are located 0.5 cun lateral to the spinous processes from T1 to L5 and are anatomically close to the paraspinal muscles and posterior nerve roots. Stimulation of these points may modulate pain pathways and improve lumbar function.

This study is designed as a randomized controlled trial comparing TEA at EX-B2 points with sham TEA in patients with chronic low back pain. The primary outcome is change in disability measured by the Oswestry Disability Index (ODI) at weeks 2, 4, 6, and 8 after intervention. The secondary outcome is change in lumbar flexibility measured by Finger-to-Floor Distance (FFD) at weeks 4 and 8. Adverse events related to the procedure will also be recorded to evaluate safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥ 18 years
* Participants experiencing low back pain for at least 3 months (>12 weeks)
* Highest low back pain intensity within the past 2 weeks with a score of ≥ 3 on a 0-10 Numeric Pain Rating Scale (NPRS)
* Receiving pharmacological therapy with a stable analgesic regimen for at least 2 weeks prior to enrollment
* Presence of physical functional disability as indicated by an Oswestry Disability Index (ODI) score > 20%
* Willing and able to participate in the study until completion and to provide written informed consent

Exclusion Criteria:

* History of hypersensitivity reactions to acupuncture or thread embedding acupuncture, or known allergy to stainless steel or polydioxanone (PDO) threads
* History of keloid formation
* Presence of scars (cicatrices) or skin disorders at the thread embedding acupuncture insertion sites in the lower back area
* Specific spinal pathology including fracture, tumor, infection, or severe lumbar spinal stenosis requiring surgical intervention
* Structural spinal abnormalities (scoliosis or kyphosis) detected on physical examination
* History of spinal surgery or indication for spinal surgery due to severe neurological deficits
* Presence of cardiac disease, hematological disorders, or uncontrolled diabetes mellitus
* Regular use of systemic steroids, nonsteroidal anti-inflammatory drugs (NSAIDs), antiplatelet agents, anticoagulants, or topical analgesic medications
* Receipt of other treatments for low back pain, including dry needling, neuromuscular taping, spinal injections, or acupuncture within the past 2 weeks, or thread embedding acupuncture within the past 6 months
* Severe cognitive impairment, severe psychiatric or psychological disorders, or history of alcohol or substance abuse
* Pregnant or breastfeeding women, or women planning pregnancy within the next 6 months
* Body mass index (BMI) < 18 kg/m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | Baseline, Week 2, Week 4, Week 6, and Week 8
  The Oswestry Disability Index (ODI) is a validated questionnaire assessing disability related to low back pain. Scores range from 0 to 100, with higher scores indicating greater disability and worse functional status. A decrease in ODI score represents improvement in functional disability.

SECONDARY OUTCOMES:
Change in Finger-to-Floor Distance (FFD) | Baseline, Week 4, and Week 8
  The Finger-to-Floor Distance (FFD) assesses lumbar flexibility by measuring the distance (in centimeters) between the fingertips and the floor during maximal forward trunk flexion. Values range from 0 cm to higher positive values, with lower scores indicating better lumbar flexibility. A decrease in FFD represents improvement in lumbar flexibility.

OTHER OUTCOMES:
Incidence and Type of Adverse Events Related to Thread Embedding Acupuncture | Through study completion, an average of 8 weeks.
  The incidence and type of adverse events related to thread embedding acupuncture will be recorded throughout the study period, including pain, bruising, swelling, infection, and other procedure-related complications. The number of participants experiencing at least one adverse event and the type of events will be summarized for each study group.

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospital (HREC FMUI-CMH) (Komite Etik Penelitian Kesehatan Fakultas Kedokteran Universitas Indonesia - RSUP Nasional Dr. Cipto Mangunkusumo)
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly. Only aggregate study results will be reported in publications.